CLINICAL TRIAL: NCT07192861
Title: Beta-cell Evaluation Through Data-driven Assessments (BETA): Pilot Study in Type 1 Diabetes
Brief Title: BETA - Pilot Study
Status: Enrolling by invitation | Type: Observational
Sponsor: 4YouandMe (Other)
Collaborators: Buck Institute for Research on Aging (Other); Phenome Health (Unknown)
Responsible Party: Principal Investigator, Stephen Friend, President, 4YouandMe
Other Study IDs: 4UBETAPILOT
Record Dates: First submitted 2025-09-18; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Diabetes (DM)
Keywords: wearables; Diabetes; smartphone app; lifestyle; stress; CGM
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frequently sampled Oral Glucose Tolerance Test (OGTT) with glucose, insulin and C-peptide at each time point; fasting HbA1c and lipid profile
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is testing the feasibility of using non-invasive, remote digital tools including continuous glucose monitors (CGMs) and Oura ring and the Empatica EmbracePlus smart wristband to predict the function of beta-cells, the cells in the pancreas that secrete insulin. This study is being initially done with individuals with Type 1 diabetes, so that in the future these methods can be tested in a larger study of individuals with Type 2 diabetes or prediabetics. The eventual aim of this work is to develop remote digital tools that can predict the health and functioning of the pancreas in people with prediabetes and Type 2 diabetes, allowing personalized treatment approaches to preserve insulin secretion.

DETAILED DESCRIPTION:
The ultimate objective of our research program is to construct a real-time, non-invasive predictor of pancreatic beta-cell function for individuals with T2D or prediabetes, using data from a CGM alongside a rich tapestry of health, lifestyle, and behavioral metrics gathered via a smartphone and a smartwatch. In the current pilot study, we will study individuals with Type 1 diabetes (T1D) who have minimal beta-cell function, to assess the feasibility of our methods for application in a subsequent, larger study of individuals with T2D or prediabetes.

To establish a robust foundation for our predictive model, 28 study participants will undergo detailed evaluations of pancreatic beta-cell function at the Buck Institute's Clinical Research Unit (CRU) using the Minimal Model Oral Glucose Tolerance Test (OGTT) with analysis of C-peptide, glucose, and insulin levels. Participants will also wear and use their own CGM, and will be provided with an Oura ring and Empatica EmbracePlus wristband to wear for up to 6 months. Participants will complete 6 at-home remote stress and meal challenges. From this data, we can calculate clinical measures of beta-cell function, including oral Disposition Index as well as measures of the Homeostatic Model Assessment of beta-cell function (HOMA-B), and beta-cell glucose sensitivity.

This hybrid approach, blending advanced digital data acquisition with traditional clinical assessments, will facilitate the identification of critical data patterns and biomarkers correlating with beta-cell function. The envisioned outcome is a powerful, scalable tool for the early identification of individuals experiencing a decline in beta-cell function.

Coalition and Collaboration partners This project is done by 4YouandMe in collaboration with The Buck Institute, Phenome Health, AgileOps, and Vector Institute and is funded by ARPA-H

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* An established diagnosis of Type 1 diabetes
* Self-reported glycated hemoglobin (HbA1c) below 8% (64 mmol/mol)
* Body Mass Index 18-40 kg/m2
* Fluent in written and spoken English
* Own a personal iPhone 6s or later (iOS 15+ or newer) or Android smartphone (version 12 or newer) and willing to use this phone to download and use the app for the study
* Own a personal Dexcom CGM and willing to provide the study researchers access to it's data during the study.
* Willing to use the study wearable devices (Oura ring, Empatica wristband)
* Resides in the San Francisco Bay area and willing to travel to Novato, CA on at least two occasions for the in person assessments at the Buck Institute.
* If using long-acting insulin (e.g. Basaglar, Lantus, Levemir, Toujeo, Tresiba), must be on a dosing schedule that involves administration of insulin only at bedtime and no other times of day
* Willing to stop use of prescription or over-the-counter medications containing acetaminophen (e.g. Tylenol, Percocet, Nyquil and other common medications for cold and flu, etc.) due to potential interference with the study-provided continuous glucose monitor.

Exclusion Criteria:

* Pregnant or breastfeeding
* Current tobacco use
* Allergy to dairy or soy
* History of pancreatic disease (other than diabetes) or pancreatic transplantation
* Active malignancy or chemotherapy for malignancy within the past year
* History of bariatric surgery or other gastrointestinal surgery anticipated to affect glucose metabolism, or any cause of gastroparesis
* Renal, hepatic, cardiovascular, or other systemic disease likely to interfere with glucose metabolism or study participation.
* History of severe hypoglycemia or diabetes-related ketoacidosis in the prior 6 months or >2 episodes in the past 12 months.
* Overnight hospitalization for any reason in the past 3 months.
* Current use of the following medications: Calcium channel blockers (e.g., verapamil), glucocorticoids, non-selective beta blockers (e.g., propranolol), GLP-1 receptor agonists, SGLT inhibitors, DPP-4 inhibitors, sulfonylureas, meglitinides, metformin, or thiazolidinediones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Type 1 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Retention | 6 months
  Proportion of participants retained according to study protocol
Feasibility: Adherence | 6 months
  Mean adherence to completing in-app daily study measures

SECONDARY OUTCOMES:
Continuos glucose excursions | 6 months
  Participants glucose excursions will be collected from personal CGMs. A glucose excursion is defined as a change (+/- 25mg/dl) since the last CGM reading. Associations between glucose excursions and factors relating to diet, stress, sleep and activity will be estimated.

CONTACTS AND LOCATIONS:
Locations (1):
- Buck Institute for Research on Aging, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data will be shared beyond the internal research team by 4YouandMe with external qualified researchers using an ARPA-H approved data sharing platforms such as the Synapse Data Sharing Platform at Sage Bionetworks. This data sharing will occur 1 year after the last participant has exited the study. Researchers from other institutions, and other third parties will be able to apply for access to the deidentified dataset by presenting a research study plan for analysis that has been reviewed by an IRB or ethics committee. Data released through these ARPA-H approved data sharing platforms will be stored indefinitely.
Supporting Information: Study Protocol, ICF, Analytic Code